CLINICAL TRIAL: NCT04078035
Title: Transduction of Psychological Stress Into Systematic Inflammation by Mitochondrial DNA Signaling
Brief Title: Biological Response to Brief Psychological Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anna L. Marsland, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY19020140; R01MH119336 (NIH)
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Acute Inflammatory Response to Psychological Stress

STUDY DESIGN:
Intervention Model Description: The investigators propose a crossover experimental trial examining physiological responses to a socio-evaluative speech task under laboratory conditions. Participants will be tested on two occasions separated by at least 1 month. On one occasion, participants will be exposed to the speech task. On the other occasion, participants will rest quietly for the same period of time with identical assessment in the absence of the stressor. Conditions will be counterbalanced in randomized starting order across subjects.
Who Masked: Outcomes Assessor
Masking Description: Samples of plasma and serum will be identified by participant identification number only. Technicians assessing levels of biological measures in these samples will be blind to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socio-evaluative Speech Stress, then Control (Experimental): Participants will attend two laboratory sessions. At the first session, participants will complete a socio-evaluative speech task, which is a widely used, highly effective way to investigate stress responses in a laboratory setting. Participants will prepare and deliver a brief, 3-minute speech defending themselves against an alleged transgression (e.g., running a stop sign). The speech will be delivered in front of a video camera, a mirror and an audience (the interviewer and another staff member). Participants will be told that their non-verbal behaviors are being evaluated. At the second session, participants will rest quietly for the same period as the speech task, in the absence of the stressor.
  Interventions: Behavioral: Socio-evaluative speech task; Behavioral: Control, Quiet Rest
- Control, then Socio-Evaluative Speech Stress (Experimental): Participants will attend two laboratory sessions. At the first session, participants will rest quietly for 5 minutes. At the second session, participants will complete a socio-evaluative speech task, which is a widely used, highly effective way to investigate stress responses in a laboratory setting. Participants will prepare and deliver a brief, 3-minute speech defending themselves against an alleged transgression (e.g., running a stop sign). The speech will be delivered in front of a video camera, a mirror and an audience (the interviewer and another staff member). Participants will be told that their non-verbal behaviors are being evaluated.
  Interventions: Behavioral: Socio-evaluative speech task; Behavioral: Control, Quiet Rest

INTERVENTIONS:
Behavioral: Socio-evaluative speech task — 5-minute speech task designed to induce physiological arousal in a laboratory setting.
Behavioral: Control, Quiet Rest — 5-minute quiet rest period.

SUMMARY:
The investigators plan to conduct a crossover experimental trial examining physiological responses to a socio-evaluative speech task under laboratory conditions. Participants will attend two laboratory sessions. At one session participants will take part in a brief laboratory stress task and at the other participants will rest for the same period. Measures of cardiovascular response will be assessed at both sessions. In addition, blood will be drawn at multiple time points across a 125 minute period to assess changes in circulating levels of cortisol, catecholamines, markers of inflammation and cell free mitochondrial DNA in response to the task. The investigators expect that the stress task will induce a specific increase in ccf-mtDNA, which will statistically mediate subsequent peak circulating Interleukin-6 and Tumor Necrosis Factor-α levels. In secondary analyses, the investigators will examine whether stress-induced increases in circulating cortisol, epinephrine, and norepinephrine levels correlate with increases in ccf-mtDNA. These studies will establish the kinetics and magnitude of psychological stress-induced ccf-mtDNA release, the association with early stress mediators, and whether ccf-mtDNA mediates the inflammatory response to acute stress in humans.

DETAILED DESCRIPTION:
The proposed study will examine physiologic responses to acute psychological challenge in the laboratory among healthy adults. It is widely accepted that there is an increase in circulating markers of inflammation following a single bout of laboratory stress. This increase in systemic inflammation is believed to contribute to the damaging health effect of psychological stress. However, to date, the biological mechanisms by which psychological stress is transduced into inflammation are unclear. The investigators' preliminary evidence suggests that mitochondrion may play a role, with stress-induced increases in circulating levels of mitochondria- derived signaling molecules that are known to modulate immune cell function and the production of pro-inflammatory cytokines.

To test this possibility, the investigators plan to conduct a crossover experimental trial examining physiological responses to an evaluative speech task under laboratory conditions. The investigators have previously used this task to induce physiological arousal. The investigators plan to recruit 60 non-smoking volunteers (50% female, aged 20-50 years) and test these participants on two occasions separated by at least a month. On one occasion the participants will be exposed to the speech task. On the other occasion, the participants will rest quietly for the same period. Conditions will be counterbalanced. At both visits cardiovascular responses (heart rate, blood pressure, and heart rate variability) will be assessed as measures of autonomic activation before, during and after the task period. Participants will also have an intravenous catheter inserted and blood drawn at ten time points over the two hour testing period on each occasion. Blood samples will be sent to laboratories at the University of Pittsburgh and at Columbia University for the assessment of mitochondria-derived signalling molecules, inflammatory markers, and cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Non-smokers/illicit drug users
* Blood pressure below 140/90
* Weight > 110 lbs
* BMI < 30
* Fluent in English
* Women -- regular menstrual cycles over the past 12 months (defined as 21- 35 days in length)
* Able and willing to give informed consent
* Willing to abstain from alcohol and vigorous exercise for 24 hours, from food and drinks (other than water) for 3 hours and from non-prescription medications (other than oral contraception) for 2 days before testing.
* Willing to attend two laboratory stress testing sessions, give blood though an intravenous catheter, undergo medical evaluation and complete psychosocial questionnaires.

Exclusion Criteria:

* Reported history of chronic systemic immune, metabolic or mitochondrial diseases, or chronic diseases that influence the central nervous, autonomic nervous or neuroendocrine systems, e.g., autoimmune disease, chronic infections, cardiovascular disease, diabetes, chronic kidney or liver disease, cancer treatment.
* Reported psychiatric history of schizophrenia or other psychotic illness, or mood disorder.
* Resting blood pressure > 140/90 mmHg at baseline testing.
* Weight < 110 lbs
* BMI equal to or greater than 30
* Report currently taking glucocorticoid, anti-inflammatory, anti-retroviral, immunosuppressant, insulin, antiarrhythmic, antihypertensive, oral hypoglycemic, antidepressant, benzodiazepine or prescription weight loss medications or other medications known to influence the immune, autonomic or neuroendocrine systems.
* For women - Post-menopausal or irregular menstrual cycles over the past 12 months. Report current pregnancy or lactation.
* Current smokers (defined as having smoked a cigarette in the previous 3 months).
* Current illicit drug use (defined as reported use of illicit drugs such as marijuana, cocaine or heroin in the previous 3 months).
* Not fluent in English (have used English in everyday speaking and reading for at least 10 years)
* Unable or unwilling to give informed consent
* Unwilling to abstain from alcohol and vigorous exercise for 24 hours, from food and drinks (other than water) for 3 hours and from non-prescription medications (other than oral contraception) for 2 days prior to testing.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna L Marsland, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will be shared. This includes all of the individual -participant data collected during the trial. In addition, the study protocol will be made available. The Co-Principal Investigators of the study will oversee all matters related to data management and archiving. Final research data will be deposited in the digital repository of the Inter-university Consortium for Political and Social Research (ICPSR), of which the University of Pittsburgh is a member, and which receives partial funding from the NIH.
Supporting Information: Study Protocol
Time Frame: Data will be made available within nine months to one year after the publication of results bearing on the project's specific aims. The Inter-university Consortium for Political and Social Research (ICPSR) will archive the full dataset and its documentation for the long term, supporting the data through changing technologies, new media, and data formats.
Access Criteria: All publications and presentations deriving from the final research data will include information on the location of the data and how it can be accessed, well as acknowledgement of the repository and funding source. The ICPSR has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.
URL: https://www.icpsr.umich.edu/web/pages/

REFERENCES:
- [Background] Trumpff C, Marsland AL, Basualto-Alarcon C, Martin JL, Carroll JE, Sturm G, Vincent AE, Mosharov EV, Gu Z, Kaufman BA, Picard M. Acute psychological stress increases serum circulating cell-free mitochondrial DNA. Psychoneuroendocrinology. 2019 Aug;106:268-276. doi: 10.1016/j.psyneuen.2019.03.026. Epub 2019 Mar 28. PMID 31029929
- [Background] Trumpff C, Marsland AL, Sloan RP, Kaufman BA, Picard M. Predictors of ccf-mtDNA reactivity to acute psychological stress identified using machine learning classifiers: A proof-of-concept. Psychoneuroendocrinology. 2019 Sep;107:82-92. doi: 10.1016/j.psyneuen.2019.05.001. Epub 2019 May 7. PMID 31112904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited into this study between 7/23/2020 and 12/17/2021. Healthy volunteers were recruited from advertisements places around campus and through "Pitt+Me," a registry of individuals interested in participating in research taking place at the University of Pittsburgh.
Pre-assignment Details: Participants were scheduled for a screening telephone call to determine eligibility. Eligible participants were rescreened at 1st study visit and excluded if they did not meet eligibility criteria. We also excluded individuals on whom we could not insert a functioning intravenous catheter at the first study visit.
Period: Session1
Arm/Group | Socio-evaluative Speech Stress, Then Control | Control, Then Socio-Evaluative Speech Stress
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0
Period: Session 2
Arm/Group | Socio-evaluative Speech Stress, Then Control | Control, Then Socio-Evaluative Speech Stress
Started | 36 | 36
Completed | 25 | 27
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 3 | 1
Not completed — Unable to insert IV - participant elected to withdraw | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Socio-evaluative Speech Stress, Then Control | Control, Then Socio-Evaluative Speech Stress | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32 (9) | 31 (8) | 31 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 21 | 17 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 25 | 27 | 52
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72
Body Mass Index [Mean (Standard Deviation); unit: kg/M^2] | 24.30 (4.27) | 22.61 (2.68) | 23.46 (3.64)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 113.05 (7.82) | 108.06 (10.53) | 110.78 (9.42)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 68.92 (6.58) | 65.85 (6.73) | 67.42 (6.75)

OUTCOME MEASURES:

1. Primary Outcome: Cell-free Mitochondrial DNA
Description: Serum levels of mitochondrial DNA assessed from blood samples
Time Frame: 5 minutes before task, and 5, 10, 20, 30, 45, 60, 75, 90 and 120 minutes after the task.
Measure: Mean (Standard Deviation); unit: Copies per uL
Groups:
- Socio-evaluative Speech Stress Session: Participants attended two laboratory sessions order of these sessions was counterbalanced. At one of the sessions, they completed a 5-minute socio-evaluative speech task defending themselves against an alleged transgression (e.g., running a stop sign). Outcomes in this condition include responses to this stressor.
- Control Session: Participants attended two laboratory sessions. Order of sessions was counterbalanced. Presented outcome data are for the control condition only. Participants rested quietly for the 5-minute task period.
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
Copies per uL
  5 min pre-task | 165.79 (143.01) | 405.56 (1218.33)
  5 min | 175.45 (144.03) | 164.45 (133.03)
  10 min | 414.74 (1942.78) | 296.62 (629.78)
  20 min | 153.37 (144.03) | 213.27 (511.28)
  30 min | 151.50 (124.64) | 163.41 (147.62)
  45 min | 171.53 (178.85) | 172.03 (155.38)
  60 min | 150.76 (93.06) | 215.58 (437.87)
  75 min | 183.87 (216.89) | 255.99 (549.68)
  90 min | 187.20 (202.77) | 223.99 (272.97)
  120 min | 161.19 (149.77) | 232.64 (279.89)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.86, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.00015, Standard Error of Mean 0.00088

2. Primary Outcome: Interleukin-6
Description: Plasma levels of interleukin-6
Time Frame: 5 minutes before to 5, 10, 20, 30, 45, 60, 75, 90, 120 post-task periods
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
pg/ml
  5 mins pre-task | 1.52 (1.29) | 1.40 (0.99)
  5 min | 1.76 (1.31) | 1.58 (0.94)
  10 min | 1.61 (1.24) | 1.52 (0.94)
  20 min | 2.05 (1.49) | 1.78 (1.01)
  30 min | 2.01 (1.44) | 1.85 (1.29)
  45 min | 2.30 (1.70) | 2.15 (1.32)
  60 min | 2.50 (1.76) | 2.27 (1.34)
  75 min | 3.28 (3.61) | 3.06 (2.84)
  90 min | 3.80 (3.78) | 2.91 (1.97)
  120 min | 4.50 (3.92) | 4.72 (5.31)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.74, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = 0.00022, Standard Error of Mean 0.00067

3. Primary Outcome: Tumor Necrosis Factor-alpha
Description: Plasma levels of tumor necrosis factor-alpha
Time Frame: 5 minutes before to 5, 10, 20, 30, 45, 60, 75, 90, 120 post-task periods
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
pg/ml
  5 min pre-task | 5.92 (2.21) | 6.10 (2.21)
  5 min | 6.62 (1.90) | 6.81 (2.79)
  10 min | 6.59 (1.84) | 6.28 (1.92)
  20 min | 6.70 (1.72) | 6.79 (2.76)
  30 min | 6.45 (1.82) | 6.35 (1.89)
  45 min | 6.61 (1.76) | 6.74 (2.63)
  60 min | 6.41 (1.65) | 6.52 (2.51)
  75 min | 6.58 (1.68) | 6.79 (2.64)
  90 min | 3.78 (6.68) | 6.75 (1.74)
  120 min | 3.92 (6.43) | 6.66 (2.62)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.52, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.0012, Standard Error of Mean 0.0019

4. Secondary Outcome: Heart Rate
Description: Continuous measurement of heart rate was averaged across 4 periods: last 5 minutes of baseline, 5-min task-period, first two 5 minutes post-task.
Time Frame: last 5 minutes of baseline, 5-min task-period, first two 5 minutes post-task.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
Beats per minute
  Mean of 5 min pre-task | 65.60 (9.57) | 66.76 (9.53)
  mean of 5 min task period | 79.27 (14.44) | 66.36 (9.46)
  mean of min 1-5 post-task | 71.37 (10.83) | 67.43 (9.20)
  mean of min 6-10 post-task | 66.00 (9.46) | 65.03 (9.24)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Test type: Superiority — Results present the condition (stress/control) by time^2 interactions; p < .001, Mixed Models Analysis; Likelihood ratio test showed better fit if quadratic for time included χ2 (2) = 77.2, p < .001; Slope = -.34, Standard Error of Mean 0.04

5. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was assessed twice on 10 occasions across the protocol. The two readings on each occasion were averaged.
Time Frame: 5 min pre-task and 5, 10, 20, 30, 45, 60, 75, 90, 120
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
mmHg
  5 min pre-task | 111.18 (9.47) | 109.43 (10.18)
  5 min post-task | 120.29 (11.71) | 110.70 (9.46)
  10 min post-task | 120.02 (12.58) | 109.38 (9.95)
  20 min post-task | 131.55 (18.09) | 109.23 (10.43)
  30 min post-task | 135.63 (16.62) | 108.98 (10.15)
  45 min post-task | 133.42 (14.32) | 109.14 (10.12)
  60 min post-task | 125.43 (13.54) | 109.46 (10.59)
  75 min post-task | 120.61 (12.45) | 109.59 (12.07)
  90 min post-task | 117.15 (10.58) | 109.29 (10.12)
  120 min post-tsk | 115.45 (12.59) | 108.32 (12.25)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results-interaction between time2 and condition; Test type: Superiority; p < .001, Mixed Models Analysis; Likelihood ratio test showed better fit if quadratic for time included χ2 (2) = 66.4, p < .001; Slope = 0.0021, Standard Error of Mean 0.00027

6. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure was assessed two times on 10 occasions across the protocol. On each occasion, the two measures were averaged.
Time Frame: 5 min pre-task and 5, 10, 20, 30, 45, 60, 75, 90, 120 post task onset
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
mmHg
  5 min pre-task | 67.69 (9.47) | 65.74 (10.18)
  5 min post-task onset | 72.00 (11.71) | 66.02 (9.46)
  10 min post task onset | 72.65 (12.58) | 65.17 (9.95)
  20 min post task onset | 79.58 (18.09) | 65.27 (10.43)
  30 min post task onset | 81.57 (16.62) | 66.42 (10.15)
  45 min post task onset | 79.03 (14.32) | 65.71 (10.12)
  60 min post task onset | 71.80 (13.54) | 66.17 (10.59)
  75 min post task onset | 68.02 (12.45) | 65.86 (12.07)
  90 min post task onset | 66.37 (10.58) | 64.34 (10.12)
  120 min post task onset | 66.30 (12.59) | 64.10 (12.25)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results-interaction between time^2 and condition; Test type: Superiority; p < .001, Mixed Models Analysis; Likelihood ratio test showed better fit if quadratic for time included χ2 (2) = 77.2, p < .001; Slope = 0.0013, Standard Error of Mean 0.0002

7. Secondary Outcome: Cortisol
Description: Circulating levels of cortisol assessed by ELISA
Time Frame: 5 minutes before to 10, 20, 30, 45, 60 minutes post-task periods
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
ug/dL
  5 min pre-task | 1.50 (0.72) | 1.48 (0.76)
  10 min post task onset | 1.46 (0.76) | 1.30 (0.62)
  20 min post task onset | 1.57 (0.86) | 1.30 (0.63)
  30 min post task onset | 1.49 (0.64) | 1.24 (0.64)
  45 min post task onset | 1.43 (0.62) | 1.24 (0.66)
  60 min post task onset | 1.35 (0.72) | 1.18 (0.60)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.005, Mixed Models Analysis; Slope = 0.0037, Standard Error of Mean 0.0013

8. Secondary Outcome: Epinephrine
Description: Levels of epinephrine in plasma
Time Frame: 5 minutes before to 5, 10, 20, 30, & 60 minutes post-task periods
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
pg/ml
  5 min pre-task | 50.56 (20.09) | 48.62 (21.67)
  5 min post task onset | 54.01 (23.87) | 47.46 (21.19)
  10 min post task onset | 49.81 (18.69) | 52.48 (28.98)
  20 min post task onset | 47.95 (18.12) | 45.16 (17.38)
  30 min post task onset | 47.08 (16.63) | 44.26 (18.35)
  60 min post task onset | 48.34 (17.78) | 41.64 (16.43)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.92, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.0071, Standard Error of Mean 0.074

9. Secondary Outcome: Norepinephrine
Description: Levels of norepinephrine in plasma
Time Frame: 5 minutes before to 5, 10, 20, 30, & 60 minutes post-task periods
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
pg/ml
  5 min pre-task | 522.86 (228.82) | 480.48 (175.92)
  5 min post-task onset | 540.39 (178.62) | 485.44 (157.60)
  10 min post-task | 526.93 (187.47) | 484.38 (151.81)
  20 min post-task | 494.17 (173.34) | 470.70 (172.50)
  30 min post-task | 477.84 (191.16) | 476.14 (155.51)
  60 min post-task | 472.74 (156.83) | 461.97 (160.05)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.04, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.85, Standard Error of Mean 0.41

10. Secondary Outcome: Heart Rate Variability
Description: Interbeat intervals of heart rate assessed by 3-lead EKG. Measures were taken continuously from 5 minutes before the task to 10 minutes after the task. Rsults were then averaged across 4 periods: 5 minutes prior to the task, the 5-minute task period, and 5-, and 10-minutes post task
Time Frame: Pre-task, task, and 1-5 and 6-10 minutes post task
Measure: Mean (Standard Deviation); unit: log normal milliseconds
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
log normal milliseconds
  Mean across 5 min pre-task | 6.50 (1.05) | 6.58 (0.81)
  Mean across 5 min task period | 5.94 (0.96) | 6.50 (0.92)
  Mean across minutes 1-5 post-task | 6.18 (0.97) | 6.37 (0.85)
  Mean across 6-10 minutes post-task | 6.30 (0.93) | 6.43 (0.91)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results-interaction between time^2 and condition; Test type: Superiority; p = 0.002, Mixed Models Analysis — Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Likelihood ratio test showed better fit if quadratic for time included χ2 (2) = 15.64, p < .001; Slope = 0.01, Standard Error of Mean 0.0033

11. Secondary Outcome: Fatigue
Description: Momentary assessment of fatigue, measured as score on the fatigue subscale on the brief Profile of Mood States questionnaire. Scores range from 0 - 20, with higher scores reflecting more fatigue.
Time Frame: 2 minutes before and 2, 60, and 120 minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on scale
  Pre-task | 4.76 (4.02) | 5.47 (3.72)
  post-task | 2.59 (2.75) | 5.36 (3.86)
  60 min post task onset | 5.79 (4.15) | 6.48 (4.62)
  120 min post task onset | 5.50 (4.50) | 5.41 (4.36)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results _condition (stress/control) by time interactions; Test type: Superiority; p = 0.008, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = 0.014, Standard Error of Mean 0.0053

12. Secondary Outcome: Anger
Description: Momentary assessment of anger, measured as score on the anger subscale on the brief Profile of Mood States questionnaire in response to the task periods. Scores range from 0 - 12, with higher scores reflecting more anger.
Time Frame: 2 minutes before and 2-, 60-, and 120-minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on a scale
  Pre-task | 0.30 (1.03) | 0.08 (0.42)
  2 min post-task | 0.70 (1.57) | 0.20 (1.05)
  60 min post task onset | 0.49 (1.39) | 0.16 (0.72)
  120 min post task onset | 0.45 (1.51) | 0.14 (0.59)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.83, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.0003, Standard Error of Mean 0.0014

13. Secondary Outcome: Anxious Mood
Description: Momentary assessment of anxious mood, measured as score on the anxiety subscale on the brief Profile of Mood States questionnaire in response to the task periods. Scores range from 0 - 16, with higher scores reflecting more anxious mood.
Time Frame: 2 minutes before and 2-, 60- and 120-minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on a scale
  2 min pre-task | 1.44 (2.13) | 1.35 (1.97)
  2 min post-task | 3.21 (2.78) | 0.93 (1.97)
  60 min post task onset | 1.56 (2.21) | 1.24 (2.30)
  120 min post task onset | 1.29 (2.18) | 1.02 (2.46)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.03, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.0074, Standard Error of Mean 0.0033

14. Secondary Outcome: Depressed Mood
Description: Momentary assessment of depressed mood, measured as score on the depression subscale on the brief Profile of Mood States questionnaire in response to the task periods. Scores range from 0 - 12, with higher scores reflecting more depressed mood.
Time Frame: 2 minutes before and 2-, 60- and 120-minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on a scale
  2 min pre-task | 0.32 (0.91) | 0.23 (0.79)
  2 min post-task | 0.46 (1.20) | 0.27 (0.94)
  60 min post task onset | 0.64 (1.34) | 0.29 (0.94)
  120 min post task onset | 0.41 (1.12) | 0.25 (0.88)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.51, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = 0.00075, Standard Error of Mean 0.00012

15. Secondary Outcome: Vigor
Description: Momentary assessment of vigor, measured as score on the vigor subscale on the brief Profile of Mood States questionnaire in response to the task periods. Scores range from 0 - 12, with higher scores reflecting more vigor.
Time Frame: 2 minutes before and 2-, 60-, and 120-minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on a scale
  2 min pre-task | 1.84 (1.97) | 1.65 (1.87)
  2 min post-task | 3.19 (2.28) | 1.54 (1.81)
  60 min post task onset | 1.39 (1.89) | 1.03 (1.53)
  120 min post task onset | 1.91 (2.30) | 1.66 (2.09)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.04, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = -0.0053, Standard Error of Mean 0.0026

16. Secondary Outcome: Wellbeing
Description: Momentary assessment of wellbeing, measured as score on the wellbeing subscale on the brief Profile of Mood States questionnaire in response to the task periods. Scores range from 0 - 12, with higher scores reflecting more wellbeing.
Time Frame: 2 minutes before and 2-, 60- and 120-minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on a scale
  2 min pre-task | 4.25 (2.11) | 4.10 (2.04)
  2 min post-task | 3.56 (2.19) | 3.93 (2.34)
  60-min post-task | 3.61 (2.36) | 3.81 (2.31)
  120-min post-task | 3.93 (2.70) | 3.82 (2.52)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.49, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = 0.0018, Standard Error of Mean 0.0027

17. Secondary Outcome: Calm Mood
Description: Momentary assessment of calm mood, measured as score on the calm subscale on the brief Profile of Mood States questionnaire in response to the task periods. Scores range from 0 - 16, with higher scores reflecting more calm mood.
Time Frame: 2 minutes before and 2-, 60-, and 120-minutes post-task periods
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
Number analyzed (Participants) | 63 | 61
score on a scale
  2 min pre-task | 9.09 (2.85) | 9.38 (2.90)
  2 min post-task | 5.87 (2.84) | 8.83 (3.39)
  60- min post task onset | 7.59 (3.40) | 8.29 (2.91)
  120 min post task onset | 7.68 (3.18) | 7.63 (3.50)
Statistical Analysis 1: Comparison: Socio-evaluative Speech Stress Session vs Control Session; Results below present the condition (stress/control) by time interactions; Test type: Superiority; p = 0.002, Mixed Models Analysis; Subject, day (nested within subject), and time as random effects and condition (stress/control) as fixed effects; Slope = 0.013, Standard Error of Mean 0.0044

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Socio-evaluative Speech Stress Session | Control Session
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/61
Other Adverse Events (participants affected / at risk) | 0/63 | 0/61

LIMITATIONS AND CAVEATS:
The trial was disrupted by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT04078035/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT04078035/SAP_003.pdf
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04078035/ICF_001.pdf